CLINICAL TRIAL: NCT05148442
Title: A Phase Ia/Ib Study Evaluating the Safety, Tolerability and Preliminary Efficacy of IBI322 in Subjects With Myeloid Tumor
Brief Title: A Study Evaluating the Safety, Tolerability and Preliminary Efficacy of IBI322 in Subjects With Myeloid Tumor
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to the company's development strategy adjustment]
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI322A106
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Myeloid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI322 (Experimental)
  Interventions: Drug: IBI322

INTERVENTIONS:
Drug: IBI322 — Recombinant anti-human CD47/PD-L1 bispecific antibody

SUMMARY:
This is a phase I study evaluating the safety, tolerability and preliminary efficacy of IBI322 in Myeloid tumor patients.

DETAILED DESCRIPTION:
Phase 1a/1b study will be conducted to evaluate the tolerability, safety, PK, PD, immunogenicity and preliminary antitumor activity of IBI322 in patients with myeloid tumor. Phase 1a is the dose escalation part of the study and Phase 1b is the dose expansion part. Combination therapy with HMA(Azacitidine or Decitabine) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who met the diagnostic criteria of recurrent / refractory AML (WHO 2016)(primordial cells in bone marrow ≥ 5%) (excluding APL and bcr-abl positive AML ) and underwent treatment.
2. Patients who meet the diagnostic criteria of recurrent / refractory MDS (WHO 2016)and underwent treatment.
3. Patients with recurrent / refractory Essential thrombocythemia (WHO2016) after treatment (for Phase Ia)
4. Male or female subject above 18 years old
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) performance status 0 ~ 2.
6. Must have adequate organ function

Exclusion Criteria:

1. Previous history with myeloproliferative Neoplasms(MPN) or MDS/MPN
2. Transformation or treatment related AML/MDS.
3. PV/MF/AML/MDS evolved from Essential thrombocythemia
4. Relapse after allogeneic hematopoietic stem cell transplantation, or autologous hematopoietic stem cell transplantation within 1 year
5. Central nervous system leukemia infiltration
6. Previous history of chronic hemolytic anemia or screening Coombe test positive
7. Previous exposure to any anti-CD47 monoclonal antibody, SIRPα antibody, or CD47/SIRPα recombinant protein.
8. Previous exposure to chimeric antigen receptor T cell immunotherapy (CAR-T)
9. Patients who received immunotherapy, targeted therapy, biological therapy or any clinical research treatment within 14 days before receiving the first dose
10. Uncontrolled concurrent diseases
11. Subjects who are allergic to the ingredients of the study drug
12. Subjects who have used immunosuppressive drugs within 7 days before the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Number of treatment related AEs | Up to 90 days post last dose
  safety and tolerability

SECONDARY OUTCOMES:
Number of patients with response | Last patient enrolled+24 weeks
  preliminary efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of soochow university, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No